CLINICAL TRIAL: NCT01406314
Title: A Phase 1, Open Label, Dose Characteristic Study to Investigate the Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of Intravenous and Subcutaneous Doses of GSK2315698A in Patients With Systemic Amyloidosis
Brief Title: SAP Depleter Dose Assessment Study in Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 114527
Record Dates: First submitted 2011-07-26; First posted 2011-08-01 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Amyloidosis
Keywords: Phase 1; Patient; Systemic Amyloidosis; Amyloidosis
MeSH Terms: conditions — Amyloidosis; Immunoglobulin Light-chain Amyloidosis | interventions — miridesap

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Intravenous infusion for approximately 48 hours followed by subcutaneous injection
  Interventions: Drug: GSK2315698

INTERVENTIONS:
Drug: GSK2315698 — Intravenous infusion for approximately 48hours followed by subcutaneous injection

SUMMARY:
This study aims to provide safety information on the ligand, GSK2315698A. The pharmacokinetics and pharmacodynamics of the ligand will be determined together with the differences in routes of dose administration, namely the tolerability between intravenous versus subcutaneous dose administration. The study will be carried out in patients with systemic amyloidosis and the ability of GSK2315698A in depleting levels of serum amyloid protein (SAP) will be measured.

DETAILED DESCRIPTION:
This study is an open label, dose characteristic study assessing safety and pharmacokinetic and pharmacodynamic considerations of GSK2315698A. GSK2315698A is a ligand known to bind to serum amyloid protein (SAP), a key component of an anti-SAP approach to the treatment of systemic amyloidosis. Safety assessments will include adverse events, vital signs, ECGs and other relevant clinical laboratory tests. Dose administration routes will also be determined focusing on the tolerability of intravenous dose administration versus subcutaneous. The study aims to recruit up to 30 patients with a medical diagnosis of systemic amyloidosis. Subjects will be asked to attend 2 dosing sessions, each session will involve an intravenous infusion of GSK2315698A over 48 hours followed by a single subcutaneous dose in session 1 and up to 3 subcutaneous doses in session 2 to be administered over a 24 hour period.

ELIGIBILITY:
Inclusion Criteria:

* medically diagnosed with systemic amyloidosis
* AST,ALT, alkaline phosphatase <= 3xULN and bilirubin ,1.5xULN
* undergone radio-labelled-SAP scanning as part of their routine clinical care
* male or female between 18 and 80 years of age inclusive, at time of signing the informed consent
* subject is ambulant and capable of attending CUC
* capable of giving written consent, which includes compliance with the requirements of the requirement and restrictions listed in the consent form
* a female subjects is eligible to participate if she is of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea
* male subjects with female partners of child-bearing potential must agree to use contraception methods listed in the protocol and informed consent information. This must be followed from the time of the first dose of study medication to 85 days post-last dose.
* smokers (<10 cigarettes a day) are permitted but must be willing to abstain for the duration of residential study sessions

Exclusion Criteria:

* a positive pre-study Hepatitis B surface antigen or Hepatitis C antibody result within 3 months of screening
* the subject has participated in a clinical trial and has received an investigational therapeutic product (unlicensed) within 3 months, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer)
* pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing
* lactating females
* unwillingness or inability to follow the procedures outlined in the protocol
* subject is mentally or legally incapacitated
* renal failure requiring haemodialysis will normally result in exclusion. Subjects in patient group 4 on haemodyalysis may be considered providing their schedule of dialysis can be accommodated within the study schedule
* decompensated cardiac failure or recent history of syncope
* clinically significant anaemia - Hb<9g/dL
* use of prohibited medications
* poor or unsuitable venous access
* subjects with a QTc of > or equal to 480ms or other ECG abnormalities which, in the opinion of the investigator, is clinically significant in that they may increase safety risk
* uncontrolled hypertension with systolic BP> 170mm Hg and/or diastolic >100 mm Hg
* previous surgical procedures that result in altered anatomy of the upper digestive tract including cholecystectomy (gall bladder removal) will result in exclusion from the Entero-Test procedure, but the subject may still participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-10-13 (Actual); Primary Completion 2012-11-14 (Actual); Study Completion 2012-11-14 (Actual)

PRIMARY OUTCOMES:
Blood concentrations of SAP | 19 weeks
  comparison of predicted vs observed
Plasma concentrations of GSK2315698 | 19 weeks
  changes in plasma concentrations of GSK2315698 over time

SECONDARY OUTCOMES:
safety and tolerability of GSK2315698 | 19 weeks
  evaluated by adverse event (AE) reporting, clinical laboratory tests, vital signs, and 12-lead electrocardiogram (ECG).
Change from baseline in blood SAP levels | 19 weeks
  evaluate effect of GSK2315698 on SAP levels in the blood

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom

REFERENCES:
- See also: Results for study 114527 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/114527?search=study&study_ids=114527#rs